CLINICAL TRIAL: NCT04927117
Title: Evaluation of Binocular Visual Acuity in Myopic Cataract Patients Using Trifocal Intraocular Lens : a 2 Years Prospective, Observational, Multi-center Study
Brief Title: Evaluation of Visual Acuity in Myopic Cataract Patients Using Trifocal Intraocular Lens
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: SHAIER2021IRB02
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-03

CONDITIONS: Cataract; Myopia; Intraocular Lens
Keywords: Myopia; visual acuity; monocular defocus curve; binocular contrast sensitivity
MeSH Terms: conditions — Cataract; Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high myopic group (group1:AL≥26.0 mm): axial length≥26.0 mm)
- age-matched control group: axial length<26.0mm

SUMMARY:
The PanOptix trifocal IOL is a new trifocal intraocular lens which is proved to provide good range of vision for distance, intermediate and near and good visual quality in cataract patients with normal axial length. But whether it can get the same visual quality in myopia is still unknown

DETAILED DESCRIPTION:
There are a few publications of multi-focal IOLs on Chinese patients with high myopia. From published papers, it is known that performance of multifocal IOLs is satisfied in myopic patients. However there is no publication to investigate PanOptix in moderate and high myopic patients. So it is imperative to demonstrate good performance of PanOptix in those special patients. The purpose of this study is to assess visual performance and patient satisfaction after the implantation of PanOptix in myopic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Axial myopic patients（Refractive condition match the axial length after eliminate the nuclear cataract induced myopia factor）
2. Corneal astigmatism <1.0D (IOL-Master 500/700, Carl Zeiss Meditec, Jena, Germany);
3. Eyes with pupil diameter>2.5 mm (Photopic) and<6 mm (Mesopic) (Pentacam HR, Oculus Optikgerate GmbH);
4. Eyes with angle kappa<0.50 mm (Pentacam HR);
5. Eyes with corneal spherical aberration<0.50 (Pentacam HR)

Exclusion Criteria:

1. Irregular corneal astigmatism
2. Any retinal disease, macular disease(Including myopic MD and retinal diseases) could affect VA, glaucoma and other severe intraocular diseases
3. Moderate-severe dry eye
4. Amblyopia（BCDVA<0.7 before cataract appears）
5. Patients having difficulties with examinations or 3 months' follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Myopic Cataract Patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Axial length (AL) | 1 minute
  Measured using the partial coherence laser interferometry (IOLMaster, Carl Zeiss Meditec, Germany)
Uncorrected distance visual acuity | 10 minutes
  Uncorrected distance visual acuity (4m) were measured using the reading table model of the Early Treatment Diabetic Retinopathy Study charts (ETDRS; Vector Vision, Ltd, Greenville, OH, USA).
Uncorrected near visual acuity | 10 minutes
  Uncorrected near visual acuity (40cm) were measured using the reading table model of the Early Treatment Diabetic Retinopathy Study charts (ETDRS; Vector Vision, Ltd, Greenville, OH, USA).
Uncorrected intermediate visual acuity | 10 minutes
  Uncorrected intermediate visual acuity (60cm) were measured using the reading table model of the Early Treatment Diabetic Retinopathy Study charts (ETDRS; Vector Vision, Ltd, Greenville, OH, USA)
contrast sensitivity | 30 minutes
  Binocular contrast sensitivity was measured at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd) using the functional acuity contrast test(Test SV-1000) of the CC-100 HW 5.0 Series system

CONTACTS AND LOCATIONS:
Overall Officials: Xu Chen, Study Director — Shanghai Aier Eye Hospital China.
Locations (1):
- Xu Chen, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohnen T, Herzog M, Hemkeppler E, Schonbrunn S, De Lorenzo N, Petermann K, Bohm M. Visual Performance of a Quadrifocal (Trifocal) Intraocular Lens Following Removal of the Crystalline Lens. Am J Ophthalmol. 2017 Dec;184:52-62. doi: 10.1016/j.ajo.2017.09.016. Epub 2017 Sep 18. PMID 28923587
- [Result] Garcia-Perez JL, Gros-Otero J, Sanchez-Ramos C, Blazquez V, Contreras I. Short term visual outcomes of a new trifocal intraocular lens. BMC Ophthalmol. 2017 May 17;17(1):72. doi: 10.1186/s12886-017-0462-y. PMID 28514944
- [Result] Alio JL, Plaza-Puche AB, Alio Del Barrio JL, Amat-Peral P, Ortuno V, Yebana P, Al-Shymali O, Vega-Estrada A. Clinical outcomes with a diffractive trifocal intraocular lens. Eur J Ophthalmol. 2018 Jul;28(4):419-424. doi: 10.1177/1120672118762231. Epub 2018 Apr 5. PMID 29619883